CLINICAL TRIAL: NCT00795197
Title: A Screening Protocol to Characterize the Disease Status of Gaucher Type 1 Patients for Potential Inclusion in a Subsequent Phase 3 Clinical Study
Brief Title: A Screening Study Evaluating Disease Status of Gaucher Type I Patients
Status: Withdrawn | Type: Observational
Why Stopped: No recruitment of patients
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: GZGD02808
Record Dates: First submitted 2008-11-19; First posted 2008-11-21 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Gaucher Disease, Type 1
Keywords: Gaucher Disease,; acid B-glucosidase,; gluco cerebrosidase,; glucosylceramide,
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Biospecimen Retention: Samples Without DNA — Blood sample/Urine sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Screening Group: Screening Group

SUMMARY:
A screening study to identify and characterize the disease status of patients with Gaucher Type 1 disease for potential inclusion in a subsequent phase 3 clinical study.

DETAILED DESCRIPTION:
The primary objective of this screening study is to identify and characterize the disease status of patients with Gaucher Type 1 disease for potential inclusion in a subsequent Phase 3 clinical study which will evaluate the efficacy and safety of Genz-112638.

This will be a multi-center, multi-national screening study to assess the disease status of patients with Gaucher Type 1 disease utilizing criteria to be eligible for enrollment in a subsequent phase 3 clinical study. The assessment performed in this study are standard of care for the evaluation of symptoms of Gaucher Type 1 disease. No study drug will be administered in this screening study.

ELIGIBILITY:
Inclusion Criteria:

* The Patient (or their parent/legal guardian) is willing and able to provide written informed consent.
* The patient has the following manifestations of Gaucher Type 1 disease identified prior to screening: A. Splenomegaly, B. Hepatomegaly, C. Anemia and /or thrombocytopenia.
* The patient is 16 to 65 years of age. For patients < 18 years of age, the patient's Tanner stage should be ≥ 4.

Exclusion Criteria:

* The patient has had a partial splenectomy within 36 months prior to screening or has had a total splenectomy.
* The patient has received miglustat within 3 months prior to screening.
* The patient has received enzyme replacement therapy within 9 months prior to screening.
* The patient is known to have evidence of neurologic (e.g., peripheral neuropathy, tremors, seizures, Parkinsonism, or cognitive impairment) or pulmonary involvement (e.g., pulmonary hypertension) as related to Gaucher Type 1 disease.
* The patient is known to have documentation of new pathological bone involvement (e.g., osteonecrosis, pathological fractures, etc.) or has a bone crisis (pain with acute onset which requires immobilization of the affected area, narcotics for relief of pain, and may be accompanied by periostal elevation, increased white cell count, fever, or immobility of > 3 days) in the 12 months prior to screening , as determined by investigator.
* The patient is transfusion dependent.
* The patient has ever had any radiation treatment.
* The patient is known to have prior esophageal varices or liver infarction.
* The patient is known to have clinically significant disease, other than Gaucher Type 1 disease, including cardiovascular, renal, hepatic, gastrointestinal, pulmonary, neurologic, endocrine, metabolic, or psychiatric disease, other medical condition, or serious intercurrent illness.
* The patient is known to have any of the following: Clinically significant family history (sudden cardiac death in 1st or 2nd degree relatives), cardiac medical history (including myocardial infraction [MI] in the past year), or cardiac assessments/symptoms consistent with ischemia.
* The patient is known to have any of the following: Specific arrythmias or finding on cardiac monitoring such as severe 1st degree atrioventricular (AV) block, any 2nd or 3rd degree AV block, highly frequent or runs (3 or more) of atrial premature contractions (APC's) or premature ventricular contractions (PVC's), complete left and right as well as partial left bundle branch block, or prolonged QT interval.
* The patient has previously tested positive for the human immunodeficiency virus (HIV) antibody, Hepatitis C antibody, or Hepatitis B surface antigen.
* The patient has received an investigational product within 30 days prior to screening.
* The patient has a history of cancer, with the exception of basal cell carcinoma.
* The patient is pregnant or lactating.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Gaucher Disease Type 1
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (3):
- The Mount Sinai School of Medicine, Department of Genetics and Genomic Sciences, New York, New York, United States
- India (2):
  - Sanjay Gandhi Postgraduate Institute of Medical Sciences (SGPGI), Lucknow
  - Jaslok Hospital and Research Center, Mumbai